CLINICAL TRIAL: NCT00800202
Title: An Open Label Study to Assess the Effect of Avastin (Bevacizumab) Combined With First Line Paclitaxel-carboplatin or Second Line Tarceva (Erlotinib) on Progression-free Survival in Non-squamous Non-small Cell Lung Cancer Patients With Asymptomatic Untreated Brain Metastasis
Brief Title: A Study of Avastin (Bevacizumab) in Patients With Non-Squamous Non-Small Cell Lung Cancer With Asymptomatic Untreated Brain Metastasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML21823; 2008-006504-33
Record Dates: First submitted 2008-12-01; First posted 2008-12-02 (Estimated); Results first posted 2014-11-19 (Estimated); Last update posted 2014-11-19 (Estimated); Status verified 2014-11

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Bevacizumab; Carboplatin; Erlotinib Hydrochloride; Paclitaxel

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: bevacizumab [Avastin]; Drug: carboplatin; Drug: paclitaxel
- 2 (Experimental)
  Interventions: Drug: bevacizumab [Avastin]; Drug: erlotinib [Tarceva]

INTERVENTIONS:
Drug: bevacizumab [Avastin] — 15mg/kg iv every 3 weeks
Drug: carboplatin — AUC6 iv every 3 weeks for 6 cycles
  Arms: 1
Drug: erlotinib [Tarceva] — 150mg/day po
  Arms: 2
Drug: paclitaxel — 200mg/m2 iv every 3 weeks for 6 cycles
  Arms: 1

SUMMARY:
This study will assess the efficacy and safety of Avastin combined with first li ne paclitaxel-carboplatin (cohort 1) or second line Tarceva (cohort 2) in patien ts with non-squamous non-small cell lung cancer with asymptomatic untreated brai n metastasis. Two cohorts of patients will be studied; the first will receive Av astin 15mg/kg iv every 3 weeks combined with first line paclitaxel 200mg/m2 iv p lus carboplatin AUC6 iv every 3 weeks for a maximum of 6 cycles, and the second cohort will receive Avastin 15mg/kg iv every 3 weeks combined with second line T arceva 150mg/kg po.The anticipated time on study treatment is until disease prog ression, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age;
* stage IV non-squamous non-small cell lung cancer;
* asymptomatic, untreated brain metastasis;
* ECOG performance status 0-1.

Exclusion Criteria:

* previous treatment for brain metastasis;
* history of migraine or epilepsy;
* previous treatment with angiogenesis inhibitors;
* for cohort 2, previous first line treatment with Avastin or Tarceva;
* current or recent use of aspirin (>325mg/day) or full-dose anticoagulants or thrombolytic agent for therapeutic purposes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2009-04; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (21):
- France (21):
  - Bordeaux
  - Brest
  - Caen
  - Chartres
  - Créteil
  - Gap
  - Gleizé
  - La Tronche
  - Lille
  - Lyon
  - Marseille
  - Montpellier
  - Paris
  - Pierre-Bénite
  - Rennes
  - Saint-Herblain
  - Strasbourg
  - Toulon
  - Toulouse
  - Vandœuvre-lès-Nancy
  - Villejuif

RESULTS

PARTICIPANT FLOW:
Groups:
- Bevacizumab+Paclitaxel+Carboplatin: Participants received bevacizumab 15 milligrams per kilogram (mg/kg) intravenously (iv) every 3 weeks until progression or unacceptable toxicity along with paclitaxel 200 milligrams per square meter (mg/m^2) iv every 3 weeks for 6 cycles and carboplatin Area Under Curve (AUC) 6.0 milligrams per milliliter per minute (mg/mL/min) iv every 3 weeks for 6 cycles. Bevacizumab was used in addition to standard first line chemotherapy.
- Bevacizumab+Erlotinib: Participants received bevacizumab 15 mg/kg iv every 3 weeks until progression or unacceptable toxicity along with erlotinib150 milligrams per day (mg/day) administered as tablets orally until progression or unacceptable toxicity. Bevacizumab was used as second-line treatment in addition to erlotinib.
Period: Overall Study
Arm/Group | Bevacizumab+Paclitaxel+Carboplatin | Bevacizumab+Erlotinib
Started | 67 | 24
Completed | 0 | 0
Not Completed | 67 | 24
Not completed — Adverse Event | 7 | 6
Not completed — Death | 1 | 0
Not completed — Other | 5 | 0
Not completed — Disease Progression | 54 | 18

BASELINE CHARACTERISTICS:
Population: The Intent-to-Treat (ITT) population: All participants enrolled in each arm who had at least one post-enrollment evaluation. Participants who were lost to follow-up immediately after enrollment were not included in the ITT population.
Groups:
- Bevacizumab+Paclitaxel+Carboplatin: Participants received bevacizumab 15 mg/kg iv every 3 weeks until progression or unacceptable toxicity along with paclitaxel 200 mg/m^2 iv every 3 weeks for 6 cycles and carboplatin: AUC 6.0 mg/mL/min iv every 3 weeks for 6 cycles. Bevacizumab was used in addition to standard first line chemotherapy.
- Bevacizumab+Erlotinib: Participants received bevacizumab 15 mg/kg iv every 3 weeks until progression or unacceptable toxicity along with erlotinib 150 mg/day administered as tablets orally until progression or unacceptable toxicity. Bevacizumab was used as second-line treatment in addition to erlotinib.
- Total: Total of all reporting groups
Arm/Group | Bevacizumab+Paclitaxel+Carboplatin | Bevacizumab+Erlotinib | Total
Number analyzed (Participants) | 67 | 24 | 91
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.37 (8.31) | 54.17 (9.73) | 58.74 (9.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 13 | 34
  Male | 46 | 11 | 57

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Progression-Free Survival (PFS) Without Disease Progression or Death at 6 Months
Description: Tumor progression was defined according to Response Evaluation Criteria In Solid Tumors (RECIST) criteria version 1.1 as increase by at least 20% in the sum of the longest diameters of each target lesion, taking as a reference the smallest sum of the longest diameters, reported since the start of treatment, or appearance of one or more new lesions. PFS (investigator assessed) was defined as the time between the first dose of study treatment and the first event of progression or death by any cause. Participants without an event were censored the last time they were known to be progression free. PFS was analyzed using the Kaplan-Meier method in each treatment arm.
Time Frame: 6 months
Population: ITT Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab+Paclitaxel+Carboplatin | Bevacizumab+Erlotinib
Number analyzed (Participants) | 67 | 24
percentage of participants | 56.5 [43.8 to 67.4] | 57.2 [37.0 to 76.3]

2. Primary Outcome: Percentage of Participants With Disease Progression or Death
Description: Tumor progression was defined according to the RECIST criteria as increase by at least 20% in the sum of the longest diameters of each target lesion, taking as a reference the smallest sum of the longest diameters, reported since the start of treatment, or appearance of one or more new lesions. PFS (investigator assessed) was defined as the time between the first dose of study treatment and the first event of progression or death by any cause. Participants without an event were censored the last time they were known to be progression free. PFS was analyzed using the Kaplan-Meier method in each treatment arm.
Time Frame: Screening, Day 1 of Cycles 3 and 5 and every 2 cycles until end of treatment visit or disease progression or death up to 18 months after enrollment of last participant
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab+Paclitaxel+Carboplatin | Bevacizumab+Erlotinib
Number analyzed (Participants) | 67 | 24
percentage of participants | 89.6 | 91.7

3. Primary Outcome: Time to Disease Progression or Death
Description: Tumor progression was defined as increase by at least 20% in the sum of the longest diameters of each target lesion, taking as a reference the smallest sum of the longest diameters, reported since the start of treatment, or appearance of one or more new lesions. Time to event was determined as the number of months between the first dose of study treatment and the first event of progression or death by any cause. PFS was analyzed using the Kaplan-Meier method in each treatment arm.
Time Frame: as for outcome 2
Population: ITT Population; only participants with progression or death were included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab+Paclitaxel+Carboplatin | Bevacizumab+Erlotinib
Number analyzed (Participants) | 60 | 22
months | 6.7 [5.7 to 7.1] | 6.3 [3.0 to 8.4]

4. Secondary Outcome: Percentage of Participants Who Died
Time Frame: Day 1 of Cycles 1, 2, 3, 4, 5, 6 and every 3 weeks up to 18 months or until death
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab+Paclitaxel+Carboplatin | Bevacizumab+Erlotinib
Number analyzed (Participants) | 67 | 24
percentage of participants | 83.6 | 91.7

5. Secondary Outcome: Probability of Being Alive at 12 and 18 Months
Time Frame: Months 12 and 18
Population: ITT Population
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Bevacizumab+Paclitaxel+Carboplatin | Bevacizumab+Erlotinib
Number analyzed (Participants) | 67 | 24
percent
  12 Months | 64.2 [51.5 to 74.4] | 50.0 [30.5 to 69.5]
  18 Months | 43.3 [31.3 to 54.7] | 41.7 [23.1 to 61.5]

6. Secondary Outcome: Time to Death
Description: Time to death was determined as the number of months between the first dose of study treatment and the event of death by any cause. Overall survival was analyzed using the Kaplan-Meier method.
Time Frame: Day 1 of Cycles 1, 2, 3, 4, 5, 6 and every 3 weeks up to 18 months or until death
Population: ITT Population; only participants with an event of death were included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab+Paclitaxel+Carboplatin | Bevacizumab+Erlotinib
Number analyzed (Participants) | 56 | 22
months | 16.0 [12.0 to 21.0] | 12.0 [8.9 to 20.2]

7. Secondary Outcome: Percentage of Participants Achieving a Best Overall Response of Complete Response or Partial Response as Assessed by the Investigator Using RECIST
Description: Overall response defined as best response according to RECIST recorded from date of randomization until disease progression or recurrence. Complete Response (CR): disappearance of all target lesions; Partial response (PR): reduction by at least 30 percent (%) of sum of the longest diameters of each target lesion, taking initial sum of longest diameters as a reference. Participants with a missing response were considered non-responders. 95% CI for one sample binomial using Pearson-Clopper method.
Time Frame: as for outcome 2
Population: ITT Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab+Paclitaxel+Carboplatin | Bevacizumab+Erlotinib
Number analyzed (Participants) | 67 | 24
percentage of participants | 62.7 [50.0 to 74.2] | 12.5 [2.7 to 32.4]

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from the date of randomization until end of study or death.
Arm/Group | Bevacizumab+Paclitaxel+Carboplatin | Bevacizumab+Erlotinib
Serious Adverse Events (participants affected / at risk) | 27/67 | 7/24
Other Adverse Events (participants affected / at risk) | 67/67 | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab+Paclitaxel+Carboplatin (N=67) | Bevacizumab+Erlotinib (N=24)
Neutropenia (Blood and lymphatic system disorders) | 16 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 0
Anaemia (Blood and lymphatic system disorders) | 2 | 0
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 2 | 0
Bicytopenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
General physical health deterioration (General disorders) | 2 | 0
Hyperthermia (General disorders) | 1 | 0
Injection site extravasation (General disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 1 | 0
Epilepsy (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0
Hypertensive encephalopathy (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 1
Glomerulonephropathy (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 1
Arrhythmia (Cardiac disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Oesophageal ulcer (Gastrointestinal disorders) | 0 | 1
Portal vein thrombosis (Hepatobiliary disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Peripheral artery thrombosis (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 2
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab+Paclitaxel+Carboplatin (N=67) | Bevacizumab+Erlotinib (N=24)
Asthenia (General disorders) | 48 | 15
Mucosal inflammation (General disorders) | 9 | 5
Pyrexia (General disorders) | 9 | 3
Xerosis (General disorders) | 0 | 10
Neutropenia (Blood and lymphatic system disorders) | 33 | 0
Anaemia (Blood and lymphatic system disorders) | 23 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 23 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 3
Insomnia (Psychiatric disorders) | 0 | 3
Nausea (Gastrointestinal disorders) | 28 | 6
Constipation (Gastrointestinal disorders) | 18 | 5
Diarrhoea (Gastrointestinal disorders) | 18 | 15
Vomiting (Gastrointestinal disorders) | 17 | 6
Abdominal pain (Gastrointestinal disorders) | 0 | 3
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 3
Paraesthesia (Nervous system disorders) | 19 | 0
Neuropathy peripheral (Nervous system disorders) | 16 | 0
Headache (Nervous system disorders) | 11 | 8
Dizziness (Nervous system disorders) | 7 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 30 | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 6
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 5
Hypertension (Vascular disorders) | 35 | 8
Alopecia (Skin and subcutaneous tissue disorders) | 29 | 5
Rash (Skin and subcutaneous tissue disorders) | 0 | 4
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 3
Decreased appetite (Metabolism and nutrition disorders) | 25 | 7
Proteinuria (Renal and urinary disorders) | 14 | 8
Rhinitis (Infections and infestations) | 9 | 0
Folliculitis (Infections and infestations) | 0 | 11
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 9 | 3
Weight decreased (Investigations) | 8 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The study being conducted under this agreement is part of the overall study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the study, but after the first publication or presentation that involves the overall study. Sponsor may request that confidential information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.